CLINICAL TRIAL: NCT02469753
Title: Interest of Continuous Non-Steroidal Anti-Inflammatory Drug Treatment in Ankylosing Spondylitis Patients Treated by Anti-TNF Therapy in the Prevention of Radiographic Outcomes
Acronym: STOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2014/36
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Ankylosing Spondylitis
Keywords: NSAIDs; Anti-TNF; syndesmophytes; mSASSS
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients treated with anti-TNF and continuous daily NSAIDs (Experimental)
  Interventions: Drug: NSAIDs; Drug: anti-TNF
- Patients treated with anti-TNF and NSAIDs on demand (Active Comparator)
  Interventions: Drug: NSAIDs; Drug: anti-TNF

INTERVENTIONS:
Drug: NSAIDs — continuous daily
  Arms: Patients treated with anti-TNF and continuous daily NSAIDs
Drug: NSAIDs — on demand
  Arms: Patients treated with anti-TNF and NSAIDs on demand
Drug: anti-TNF

SUMMARY:
Ankylosing spondylitis (AS) is a frequent chronic inflammatory rheumatic disease that affects the axial skeleton, starting in the sacroiliac joints and spreading to the spine in most patients. Non-steroidal anti-inflammatory drugs (NSAIDs) are the primary treatment for AS. Even if the use of anti-TNF agents has demonstrated good clinical efficacy in controlling inflammation, in contrast to other conditions such as rheumatoid arthritis and psoriatic arthritis, anti-TNF treatment has failed to demonstrate any benefit on the structural progression of AS, some data even suggesting that it may accelerate the formation of syndesmophytes that seems to be an independent process of TNF. Conversely, NSAIDs inhibit ossification phenomena independently of their anti-inflammatory properties, owing to a specific action on bone formation via prostaglandin inhibition.

Several features suggest that a continuous NSAID therapy is needed, in addition to anti-TNF treatment, to prevent syndesmophyte formation in AS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* Patients who fulfil 1984 modified New York criteria for ankylosing spondylitis:
* SA patients with indications for anti-TNF treatment initiation according to the French society of Rheumatology guidelines.
* Being affiliated to a health insurance system
* Having signed an informed consent form (later than the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Patients who present another chronic systemic inflammatory disorder, different from ankylosing spondylitis.
* Patients who present contraindications to treatment with NSAIDs.
* Patient with daily corticosteroid treatment at a dosage ≥ 10 mg/day
* Pregnant or breastfeeding women
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing to undergo MRI
* Women that refuse to an effective contraception method for all the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who show a significant radiographic progression between the two randomised groups of patients | 24 month after the begin of the treatment

SECONDARY OUTCOMES:
Radiologic evolution between-group comparison | At the inclusion (Day 0) and 24 month after after the inclusion (Day 0)(begin of the treatment)
  This measure is a composite with :
  * MRI
  * Clinical evolution of patients
  * Quantitative analysis of mSASSS score

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe THIEBAUT, Prof, Study Chair — University Hospital Bordeaux, France; Thierry SCHAEVERBEKE, Prof, Principal Investigator — University Hospital Bordeaux, France
Locations (22):
- France (21):
  - Service de rhumatologie - CHU d'Amiens, Amiens
  - Service de rhumatologie - CHU de Besançon, Besançon
  - Service de Rhumatologie - CHU de Bordeaux, Bordeaux
  - service de rhumatologie - AP-HP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Service de rhumatologie - CHU de Brest, Brest
  - service de rhumatologie - CH de Cahors, Cahors
  - service de rhumatologie - CH Le Mans, Le Mans
  - service de rhumatologie - CHU de Limoges, Limoges
  - service de rhumatologie - CHU de Montpellier, Montpellier
  - service de rhumatologie - CHU de Nancy, Nancy
  - Service de rhumatologie - CHU de Nice, Nice
  - service de rhumatologie - CHR d'Orléans, Orléans
  - service de rhumatologie - AP-HP - Hôpital Henri Mondor, Paris
  - Service de rhumatologie - AP-HP - Hôpital Lariboisière, Paris
  - service de rhumatologie - AP-HP- Hôpital La Pitié Salpétrière, Paris
  - service de rhumatologuie - CH de Pau, Pau
  - service de rhumatologie - CHU de Rouen, Rouen
  - service de rhumatologie - CHU de Saint-Etienne, Saint-Etienne
  - service de rhumatologie - CHU de Strasbourg, Strasbourg
  - service de rhumatologie - CHU de Toulouse, Toulouse
  - Service de rhumatologie - CHU de Tours, Tours
- service de Rhumatologie - CH Princesse Grace, Monaco, Monaco